CLINICAL TRIAL: NCT02744482
Title: Efficacy of Risedronate in Patients With Painful Periprosthetic Resorption of the Hip Prothesis Double-blind Randomized Study Versus Placebo
Brief Title: Efficacy of Risedronate in Patients With Painful Periprosthetic Resorption of the Hip Prothesis
Acronym: PTH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of patients
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I14005
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Prosthesis Loosening
MeSH Terms: conditions — Prosthesis Failure | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risedronate (Experimental): Patients take an oral tablet of Risedronate 75 mg, 2 consecutive days per month during 18 months.
  Interventions: Drug: risedronate
- Placebo (Placebo Comparator): Patients take an oral tablet of Placebo, 2 consecutive days per month during 18 months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: risedronate — risedrante tablet (75 mg)
  Arms: Risedronate
Drug: placebo — risedrante placebo tablet (75 mg)
  Arms: Placebo

SUMMARY:
This is an experimental study, prospective, comparative. This clinical trial is randomized and double-blind, Residronate versus placebo.

The study aims to demonstrate the effectiveness of risedronate in pain management, after 18 month of traitment, in patients undergoing aseptic joint prosthesis loosening. 2 groups were compared with a 1: 1 ratio. The first group receives active drug (risedronate 75mg) and the second a placebo.

Patients are treated during 18 months: 1 tablet residronate/placebo per os two consecutive days each month.

Evaluations are planned evry 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older.
* Written informed consent
* Subjects with cemented or not cemented total hip prothesis (for primitive or secondary coxarthrosis)
* Painful aseptic loosening
* Subject has pain 4 or greater on a 10 point Visual Pain Rating scale
* For subject woman of reproductive age, they must use reliable method(s) of contraception and/or abstinence, for the duration of therapeutic product exposure.

Exclusion Criteria:

* Subjects with septic loosening of hip prosthesis

  . Subjects with bilateral disease
* Subjects with implant mobility associated with pre-operative and intraoperative loosening
* Subjects under anti-osteoporotic treatment
* Subjects having stopped a biphosphonate traetment for less than one year
* Subjects with known allergy or sensitivity to any of the components in the study medication.

  * Subjects with Hypocalcemia
  * Females who are pregnant, breast-feeding, or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
  * Subjects with severe kidney failure ( creatinine < 30 ml/min)).
  * Subjects participation in another research study
  * Subjects with previous osteonecrosis of the jaw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05; Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Pain measurement | 18, months
  Measurement of pain by means of numerical rating scale.

SECONDARY OUTCOMES:
Pain measurement at walk | 6 months, 12 months, 18, months, 24 moths
  Measurement of pain by means of numerical rating scale
Pain measurement at rest | 6 months, 12 months, 18, months, 24 moths
  Measurement of pain by means of numerical rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No